CLINICAL TRIAL: NCT02910284
Title: A Long-term Follow-up Study of Efficacy and Immunogenicity of GEN-003 in Subjects With Genital Herpes Simplex Virus Type 2 (HSV-2) Infection
Brief Title: Long-term Follow-up of GEN-003-002 Subjects for Efficacy and Immunogenicity
Status: Completed | Type: Observational
Sponsor: Genocea Biosciences, Inc. (Industry)
Responsible Party: Sponsor
Other Study IDs: GEN-003-002b
Record Dates: First submitted 2016-09-09; First posted 2016-09-22 (Estimated); Last update posted 2017-10-20 (Actual); Status verified 2017-10

CONDITIONS: Genital Herpes Simplex Type 2
Keywords: HSV; Herpes; Genital Herpes
MeSH Terms: conditions — Herpes Simplex; Herpes Genitalis | interventions — Watchful Waiting

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Biological: Observational

SUMMARY:
This study is a follow-up study from Study GEN-003-002 to evaluate long-term efficacy and immunogenicity of GEN-003 in subjects with genital HSV-2 infection.

ELIGIBILITY:
Inclusion Criteria:

1. Completion of Study GEN-003-002
2. Receipt of at least 1 dose of GEN-003 (any dose combination) in Study GEN-003-002.
3. Collection of at least 45 of 56 anogenital swabs during the Month 11 to 12 swab collection period in Study GEN-003-002.
4. Willing and able to provide written informed consent.
5. Willing to perform and comply with all study procedures, including attending clinic visits as scheduled.
6. For each swab collection period, willing to not use HSV-2 antiviral therapy from 14 days before the swab collection period through the end of the period.

Exclusion Criteria:

1. Any important protocol deviation in Study GEN-003-002.
2. Use of HSV-2 antiviral therapy within 14 days before the beginning of Swab Collection Period 1.
3. Use of topical steroids or antiviral medication in the anogenital region within 14 days before the beginning of Swab Collection Period 1.
4. Use of tenofovir, lysine, or other medication or supplement known or purported to affect HSV outbreak frequency or intensity within 14 days before the beginning of Swab Collection Period 1.
5. Immunocompromised individuals, including those receiving immunosuppressive doses of corticosteroids (more than 20 mg of prednisone given daily or on alternative days for 2 weeks or more within 6 months before the Visit 1, any dose of corticosteroids within 30 days before Visit 1, or high-dose inhaled corticosteroids [>960 µg/day of beclomethasone diproprionate or equivalent]) or other immunosuppressive agents.
6. Presence or history of autoimmune disease, regardless of current treatment.
7. Receipt of a vaccine containing HSV-2 antigens other than GEN-003.
8. Pregnant women.
9. History of drug or alcohol abuse that, in the opinion of the Investigator, would interfere with the patient's ability to comply with the requirements of the study.
10. Onset of an AESI since Month 12 in study GEN-003-002.
11. Other active, uncontrolled comorbidities that, in the opinion of the Investigator, would make the subject unsuitable for the study or unable to comply with the study requirements.

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Study Population: Subjects who received at least 1 dose of active GEN-003 and completed the GEN-003-002 study.
Sampling Method: Non-Probability Sample
Enrollment: 140 (Actual)
Dates: Start 2016-09-16 (Actual); Primary Completion 2017-07-14 (Actual); Study Completion 2017-07-14 (Actual)

PRIMARY OUTCOMES:
Long-term effect of GEN-003 on anogenital Herpes simplex virus type 2 (HSV-2) shedding (percent of anogenital swabs positive for HSV-2 DNA by PCR) | Up to 48 months post-dose
Long-term effect of GEN-003 on anogenital Herpes simplex virus type 2 (HSV-2) shedding (magnitude of HSV-2 viral shedding by PCR) | Up to 48 months post-dose

SECONDARY OUTCOMES:
Long-term effect of GEN-003 on HSV-lesion rate (percent of days with genital lesions present) during the swab collection periods | Up to 48 months post-dose
Long-term immune responses to GEN-003 (Serum IgG levels assessed by ELISA) | Up to 48 months post-dose
Long-term immune responses to GEN-003 (Serum HSV-2 neutralizing antibody levels assessed by a colorimetric neutralization assay) | Up to 48 months post-dose
Long-term immune responses to GEN-003 (Spot-forming units (SFUs), fold rise, responder rate assessed by GrB ELISPOT) | Up to 48 months post-dose

CONTACTS AND LOCATIONS:
Locations (13):
- United States (13):
  - University of Alabama - Birmingham, Birmingham, Alabama
  - Medical Center for Clinical Research, San Diego, California
  - Quest Clinical Research, San Francisco, California
  - University of Illinois - Chicago, Chicago, Illinois
  - Indiana University, Indianapolis, Indiana
  - The Fenway Institute, Boston, Massachusetts
  - University of North Carolina, Chapel Hill, North Carolina
  - Cincinnati Children's Hospital Medical Center, Cincinnati, Ohio
  - NW Dermatology and Research, Portland, Oregon
  - Magee - Women's Hospital of UPMC, Pittsburgh, Pennsylvania
  - Tekton Research, Austin, Texas
  - Center for Clinical Studies, Houston, Texas
  - University of Washington, Seattle, Washington

IPD SHARING:
Plan to Share IPD: Undecided